CLINICAL TRIAL: NCT06349291
Title: Venous Thrombosis After Removal of Central Venous Catheter-prospective Observational Study
Brief Title: Venous Thrombosis After Removal of Central Venous Catheter
Status: Recruiting | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, sara dichtwald, Dr, Meir Medical Center
Other Study IDs: 0074-24-MMC
Record Dates: First submitted 2024-03-31; First posted 2024-04-05 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Thrombosis, Venous
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Detection of venous thrombosis via US — Detection of venous thrombosis via US in patients after removal of central venous catheter

SUMMARY:
Insertion of intravenous catheter is a very common operation in patients in the general intensive care unit. These catheters are used for a variety of purposes - administration of inotropics/pressors, intravenous nutrition, concentrated electrolytes and performing dialysis.There are several known complications of central venous catheter insertion, such as thrombosis and pulmonary embolism. In a literature review, there are no clear data regarding the rate of intravenous thrombosis in patients after removal of a central venous catheter. These findings are often discovered randomly, when the patient undergoes imaging for a different indication. There is no recommendation for an active search for intravenous thrombi at the catheter insertion sites in these patients, and it is not entirely clear whether it is mandatory to administer anticoagulant treatment in these patients if thrombi are randomly discovered at the catheter insertion sites.

In this study, we aim to check the proportion of patients who developed thrombosis at the central catheter insertion sites after its removal, to check whether there are catheter insertion sites that are at a higher risk of developing thrombosis than other sites, and to check whether there are predictive characteristics for the development of this type of thrombosis.

ELIGIBILITY:
Inclusion Criteria: Patients who were admitted to the intensive care unit and had a central catheter inserted during their stay in the unit for any reason, and whose central catheter was removed during their stay in the general intensive care unit.

-

Exclusion Criteria:Patients whose insertion or removal of the central catheter did not occur during the hospitalization in the intensive care unit, patients who were treated with full anticoagulation in the intensive care unit.

-

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were admitted to the intensive care unit and had a central catheter inserted during their stay in the unit for any reason, and whose central catheter was removed during their stay in the general intensive care unit.
  -
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Rate of DVT after removal of central venous catheter | 1-3 days after removal of central venous catheter
  Rate of DVT after removal of central venous catheter as detected by US

CONTACTS AND LOCATIONS:
Locations (1):
- Meir Medical Center, Kfar Saba, Israel

IPD SHARING:
Plan to Share IPD: No